CLINICAL TRIAL: NCT03844217
Title: Copeptin After an Oral Stimulation With Macimorelin in Healthy Volunteers - The Macicop-Study
Brief Title: Copeptin After an Oral Stimulation With Macimorelin in Healthy Volunteers
Acronym: Macicop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-02205; me18ChristCrain4
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Polyuria-polydipsia Syndrome
Keywords: Copeptin; Macimorelin; Ghrelin receptor agonist; posterior pituitary gland; polyuria-polydipsia syndrome; hypothalamo-pituitary-adrenal axis
MeSH Terms: conditions — Diabetes Insipidus | interventions — macimorelin; Weights and Measures

STUDY DESIGN:
Intervention Model Description: Prospective, proof-of concept diagnostic study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Macimorelin 0.5mg/kg body weight (Experimental): Visit 1: oral Macimorelin stimulation test with the dose of 0.5mg/kg body weight Macimorelin.
  Visit 2: After a washout-phase of 1 week, participants will undergo the oral Macimorelin stimulation test with the dose of 0.75mg/kg body weight. Study procedures are equal compared to visit 1.
  Macimorelin 0.75mg/kg body weight
  Interventions: Drug: Macimorelin 0.5mg/kg body weight; Drug: Macimorelin 0.75mg/kg body weight

INTERVENTIONS:
Drug: Macimorelin 0.5mg/kg body weight — oral Macimorelin stimulation test with the dose of 0.5mg/kg body weight Macimorelin
Drug: Macimorelin 0.75mg/kg body weight — oral Macimorelin stimulation test with the dose of 0.75mg/kg body weight Macimorelin

SUMMARY:
This study investigates stimulation of the posterior pituitary gland by oral Macimorelin (a ghrelin receptor Agonist) to be a novel diagnostic test in the polyuria-polydipsia syndrome.

DETAILED DESCRIPTION:
Copeptin measurements upon intravenous arginine stimulation discriminate patients with diabetes insipidus versus patients with primary polydipsia with a high diagnostic accuracy. An oral test would be easier to perform, causes less risks and discomfort for the patients and would require less resources in clinical practice. This study investigates stimulation of the posterior pituitary gland by oral Macimorelin (a ghrelin receptor Agonist) to be a novel diagnostic test in the polyuria-polydipsia syndrome.

ELIGIBILITY:
Inclusion Criteria:

* No medication except hormonal contraception

Exclusion Criteria:

* Body Mass Index (BMI) > 40kg/m2 or BMI < 18.5 kg/m2
* participation in a trial with investigational drugs within 30 days
* vigorous physical exercise within 24 hours before the study participation
* Alcohol intake within 24 hours before study participation
* pregnancy and breastfeeding
* Evidence of disordered drinking habits and diuresis defined as polyuria >50ml/kg body weight/24h and polydipsia >3l /24h
* a prolonged QT interval (QTc >500 ms) or concomitant treatment with drugs that prolong the QT/QTc.
* Intention to become pregnant during the course of the study
* Known allergy towards Macimorelin

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
Change in Copeptin value (pmol/l), after intake of Macimorelin of 0.5mg/kg body weight | baseline blood exam (timepoint 0) and further blood collections after 30, 45, 60, 90 and 120 minutes after baseline blood collection
  evaluate copeptin values after the intake of of a single oral-dose Macimorelin of 0.5mg/kg body weight

SECONDARY OUTCOMES:
Change in Copeptin value (pmol/l), after intake of Macimorelin of 0.75mg/kg body weight | baseline blood exam (timepoint 0) and further blood collections after 30, 45, 60, 90 and 120 minutes after baseline blood collection
  evaluate copeptin values after the intake of of a single oral-dose Macimorelin of 0.75mg/kg body weight
Change in Growth Hormone (GH) value (ng/mL) | baseline blood exam (timepoint 0) and further blood collections after 30, 45, 60, 90 and 120 minutes after baseline blood collection
  evaluate GH values after the intake of of a single oral-dose Macimorelin
Change in Insulin-like growth factor 1 (IGF-1) value (yg/mL) | baseline blood exam (timepoint 0) and further blood collections after 30, 45, 60, 90 and 120 minutes after baseline blood collection
  evaluate IGF-1 values after the intake of of a single oral-dose Macimorelin
Change in free thyroxine (fT4) value (ng/dL) | baseline blood exam (timepoint 0) and further blood collections after 30, 45, 60, 90 and 120 minutes after baseline blood collection
  evaluate fT4 values after the intake of of a single oral-dose Macimorelin
Change in Thyreotropin (TSH) value (mU/L) | baseline blood exam (timepoint 0) and further blood collections after 30, 45, 60, 90 and 120 minutes after baseline blood collection
  evaluate TSH values after the intake of of a single oral-dose Macimorelin
Change in Prolactin value (yg/L) | baseline blood exam (timepoint 0) and further blood collections after 30, 45, 60, 90 and 120 minutes after baseline blood collection
  evaluate Prolactin values after the intake of of a single oral-dose Macimorelin
Change in Cortisol value (ng/mL) | baseline blood exam (timepoint 0) and further blood collections after 30, 45, 60, 90 and 120 minutes after baseline blood collection
  evaluate Cortisol values after the intake of of a single oral-dose Macimorelin
Change in Adrenocorticotropin (ACTH) value ( pg/mL) | baseline blood exam (timepoint 0) and further blood collections after 30, 45, 60, 90 and 120 minutes after baseline blood collection
  evaluate ACTH values after the intake of of a single oral-dose Macimorelin
Change in Luteotropin (LH) value (U/L) | baseline blood exam (timepoint 0) and further blood collections after 30, 45, 60, 90 and 120 minutes after baseline blood collection
  evaluate LH values after the intake of of a single oral-dose Macimorelin
Change in Follicle-stimulating hormone value(FSH) (IU/mL) | baseline blood exam (timepoint 0) and further blood collections after 30, 45, 60, 90 and 120 minutes after baseline blood collection
  evaluate FSH values after the intake of of a single oral-dose Macimorelin

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof. Dr. MD, Principal Investigator — Endocrinology, Diabetes and Metabolism, University Hospital Basel
Locations (1):
- University Hospital Basel Endocrinology, Diabetes and Metabolism, Basel, Switzerland

REFERENCES:
- [Derived] Urwyler SA, Lustenberger S, Drummond JR, Soares BS, Vogt DR, Ammer N, Yuen KCJ, Ribeiro-Oliveira A, Christ-Crain M. Effects of oral macimorelin on copeptin and anterior pituitary hormones in healthy volunteers. Pituitary. 2021 Aug;24(4):555-563. doi: 10.1007/s11102-021-01132-9. Epub 2021 Feb 22. PMID 33615399